CLINICAL TRIAL: NCT06034106
Title: The Effect of Pomegranate (Punica Granatum L.) Peel Compress Application on Pain and Physical Function Status in Patients With Knee Osteoarthritis
Brief Title: The Effect of Pomegranate (Punica Granatum L.) Peel Compress Application on Pain and Physical Function Status
Acronym: Pomegranate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Dilek Efe Arslan, ErciyesU, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: getat51
Record Dates: First submitted 2023-08-08; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Pomegranate (P. Granatum) Peel Compress
Keywords: pain; osteoarthritis; rheumatologic diseases; physical function; stiffness; nursing
MeSH Terms: conditions — Pain; Osteoarthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pomegranate (P. granatum) peel compress group (Experimental): 36 g of pomegranate peel powder was given to the patient in a closed container. A teaspoon (approximately 2-3 g) of powder was mixed with water from the storage container and applied to the patient's knee by making a paste, and then the knee was wrapped with a bandage. It was kept for 20 minutes by placing a hot thermophore (approximately 40-45 C) on it. This application was carried out 3 days a week.
  Interventions: Behavioral: Pomegranate (Punica granatum) peel compress
- Hot compress (Placebo Comparator): In the hot compress group, the knee was wrapped with a bandage and the hot thermophor (approximately 40-45 °C) was placed on the knee. The hot thermoform was applied to the patient 3 days a week by keeping it for 20 minutes.
  Interventions: Behavioral: Pomegranate (Punica granatum) peel compress; Behavioral: Hot compress
- Control Group (No Intervention): Patients in the control group did not receive any additional intervention.

INTERVENTIONS:
Behavioral: Pomegranate (Punica granatum) peel compress — Pomegranate (Punica granatum) peel compress was applied 3 days a week for 3 weeks by turning the powder into porridge check.
  Arms: Hot compress; Pomegranate (P. granatum) peel compress group
Behavioral: Hot compress — Hot compress was applied 3 days a week for 3 weeks.
  Arms: Hot compress

SUMMARY:
Osteoarthritis is the most common type of arthritis among rheumatologic diseases. Complementary therapies are one of the effective methods for pain control. This study was planned as a randomized controlled experimental study. For this purpose, patients diagnosed with knee osteoarthritis who applied to the Orthopedics Outpatient Clinic will be included. It was calculated that the study would include at least 67 patients. The study will be collected using patient information form, descriptive characteristics form, Visual Analog Scale (VAS) and WOMAC osteoarthritis application scale. It was planned as a randomized controlled experimental study to evaluate the effect of pomegranate peel (P. granatum) compress application on pain and function status. The study was divided into 3 groups as Pomegranate (Punica granatum) peel compress, hot compress and control group. Pomegranate (Punica granatum) peel compress was applied 3 days a week for 3 weeks by turning the powder into porridge check.

DETAILED DESCRIPTION:
This randomized controlled experimental study was conducted to evaluate the effect of pomegranate (Punica granatum) peel compress application on pain, stiffness and physical function in individuals with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Visual analog scale score of 3 and above,
* those aged 45 and over,
* Diagnosed with knee OA by a physician according to the criteria of the American - Rheumatology Association (ARD),
* pain lasting at least 1 month or longer,
* not included in any physical therapy program during the research period, a
* capable of answering research questions,
* agreeing to participate in the research by giving verbal and written consent

Exclusion Criteria:

* with a defined psychiatric illness,
* having vision and hearing problems,
* diagnosed with complex disease such as malignant,
* having a wound in the application area,
* with a diagnosed vascular disease,
* the patient's other inflammatory disease such as rheumatoid arthritis, gout, fibromyalgia
* who have had serious trauma or surgery in the last 6 months,
* who have received DMARDS or intra-articular steroid injection therapy in the last 3 months

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2023-04-14 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-10-15 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | The scale was filled in the baseline
  A VAS consisting of a 10-centimeter horizontal line, anchored evenly by numbers from 0 to 10, was used to assess the patient's pain and willingness to repeat the procedure. The number 0 was identical to having no pain while the number 10 corresponded to maximal pain that can be experienced by the patient
WOMAC Osteoarthritis Index | The scale was filled in the baseline
  The WOMAC index is composed of 24 items and 3 subdimensions (pain, stiffness, and physical function). The participants are asked to rate pain (5 questions), stiffness (2 questions), and difficulties encountered in physical functioning (17 questions) during the day (24 hours). The index is a 5-point Likert-type scale, where 0 is none, 1 mild, 2 moderate, 3 severe, and 4 very severe. Pain scores range from 0e20 points, stiffness scores from 0e8 points, and difficulties in physical function scores from 0e68 points. Higher scores indicate increased pain and stiffness, impairment in physical functioning, and higher levels of physical limitation.

CONTACTS AND LOCATIONS:
Overall Officials: DİLEK EFE ARSLAN, Study Director — ERCİYES UNİVERSİTY
Locations (1):
- Dilek Efe Arslan, Kayseri, Melikgazi, Turkey (Türkiye)